CLINICAL TRIAL: NCT06720415
Title: Comparison of Oral and Intravenous Methadone for Analgesia in Cardiac Surgery
Brief Title: Oral and Intravenous Methadone for Analgesia in Cardiac Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Krishnan Ramanujan, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-006579
Record Dates: First submitted 2024-11-19; First posted 2024-12-06 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Anesthesia; Cardiac Surgery
MeSH Terms: interventions — Methadone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oral methadone, immediately prior to transport (Experimental)
  Interventions: Drug: Oral methadone, immediately prior to transport
- Intravenous methadone (Active Comparator)
  Interventions: Drug: Intravenous methadone

INTERVENTIONS:
Drug: Oral methadone, immediately prior to transport — Patients will receive 0.4mg/kg PO methadone immediately prior to transport to the operating room
  Arms: Oral methadone, immediately prior to transport
Drug: Intravenous methadone — Patients will receive 0.3mg/kg IV methadone after induction of general anesthesia
  Arms: Intravenous methadone

SUMMARY:
The purpose of this study is to compare the effects of administration of oral methadone preoperatively and intravenous methadone upon induction of general anesthesia on postoperative pain for patients undergoing elective cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

• Undergoing elective cardiac surgery as the first case of the day in an operating room

Exclusion Criteria:

* Chronic pain requiring opioid medications as an outpatient
* Opioid use disorder on medication assistance treatment
* Prolonged QTc > 500ms
* Chronic kidney disease with eGFR < 30mL/min
* Documented cirrhosis
* Intolerance to methadone
* Subsequent surgeries after index surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2025-04-14 (Actual); Primary Completion 2025-07-07 (Actual); Study Completion 2025-07-14 (Actual)

PRIMARY OUTCOMES:
Opioid Use in Morphine Milligram Equivalents 24 hours after extubation | From hospital admission for surgery to 24 hours after the patient is extubated postoperatively

SECONDARY OUTCOMES:
Opioid Use in Morphine Milligram Equivalents 48 hours after extubation | From hospital admission for surgery to 48 hours after the patient is extubated postoperatively
Opioid Use in Morphine Milligram Equivalents 72 hours after extubation | From hospital admission for surgery to 72 hours after the patient is extubated postoperatively
Pain score 6 hours after extubation | From hospital admission for surgery to 6 hours after extubation postoperatively
  Pain will be assessed using a numerical rating scale from 0-10, with 0 being no pain and 10 being the worst pain imaginable.
Pain score 12 hours after extubation | From hospital admission for surgery to 12 hours after extubation postoperatively
  Pain will be assessed using a numerical rating scale from 0-10, with 0 being no pain and 10 being the worst pain imaginable.
Pain score 24 hours after extubation | From hospital admission for surgery to 24 hours after extubation postoperatively
  Pain will be assessed using a numerical rating scale from 0-10, with 0 being no pain and 10 being the worst pain imaginable.
Pain score 48 hours after extubation | From hospital admission for surgery to 48 hours after extubation postoperatively
  Pain will be assessed using a numerical rating scale from 0-10, with 0 being no pain and 10 being the worst pain imaginable.
Pain score 72 hours after extubation | From hospital admission for surgery to 72 hours after extubation postoperatively
  Pain will be assessed using a numerical rating scale from 0-10, with 0 being no pain and 10 being the worst pain imaginable.
Time to extubation | From the time the patient arrives in the ICU intubated until the time the patient is successfully extubated. If the patient is extubated in the operating room, this time will be 0.
  This outcome will monitor the time in minutes from when a patient arrives in the ICU to the time the breathing tube is removed (extubation).
Opioid Use in MMEs Prior to Extubation | From the time the patient arrives in the ICU intubated until the time the patient is successfully extubated. If the patient is extubated in the operating room, this time will be 0.
  This outcome will assess the need for pain medications (opioids) to make patients comfortable prior to removing the breathing tube (extubation).

CONTACTS AND LOCATIONS:
Overall Officials: Krishnan Ramanujan, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No